CLINICAL TRIAL: NCT02230969
Title: Plegridy™ (Peginterferon β-1a) Real World Effectiveness and Safety Observational Program
Brief Title: Plegridy Observational Program
Acronym: POP
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 105MS401
Record Dates: First submitted 2014-08-29; First posted 2014-09-03 (Estimated); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Relapsing Forms of Multiple Sclerosis
Keywords: peginterferon; relapsing; pegylated; Subcutaneous; Injectable; Multiple Sclerosis
MeSH Terms: conditions — Recurrence; Multiple Sclerosis | interventions — peginterferon beta-1a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- peginterferon beta-1a: Plegridy will not be supplied for this study. The study will collect data in an observational manner from participants who are prescribed Plegridy by physicians, according to the approved label in the respective country.
  Interventions: Drug: peginterferon beta-1a

INTERVENTIONS:
Drug: peginterferon beta-1a — Administered as specified in the treatment arm
  Other Names: BIIB017; PEG IFN β-1a; Plegridy; PEGylated Interferon Beta-1a

SUMMARY:
The primary objectives of the study are to determine the incidence of serious adverse events (SAEs) in participants with relapsing forms of multiple sclerosis (MS) in routine clinical practice and to assess the overall long-term clinical effectiveness of Plegridy in participants with relapsing forms of MS in routine clinical practice. The secondary objectives of this study in this study population are to describe Plegridy prescription and utilization adherence patterns in routine clinical practice; to assess the specific long-term clinical effectiveness of Plegridy in participants with relapsing forms of MS in routine clinical practice; to monitor the safety and tolerability of Plegridy in routine clinical practice by assessing the incidence of adverse events (AEs) of flu-like symptoms (FLS), injection site reactions (ISRs), and AEs (including laboratory abnormalities) leading to treatment discontinuation; to assess the effect of FLS on participant-reported effectiveness of, and satisfaction with, prophylactic management using a FLS-Visual Analog Scale (FLS-VAS); to evaluate the change in health-related quality of life (HRQoL), FLS, FLS-VAS, healthcare resource consumption, and treatment adherence over time.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient with MS who is newly, or is currently, prescribed Plegridy according to local label including patients who participated in Study 105MS302 (NCT01332019) or Study 105MS303 (NCT01939002).
* Patient willing and able to complete patient-reported outcomes (PRO) with minimal assistance.

Key Exclusion Criteria:

* Concurrent enrollment in any clinical trial of an investigational product. Participation in non-interventional study can be allowed as long as this participation does not interfere with this protocol or is likely to affect the subject's ability to comply with the protocol.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in participants with relapsing forms of MS who are newly or currently prescribed Plegridy as prescribed under routine clinical practice and participants who participated in Study 105MS302 (NCT01332019) or Study 105MS303 (NCT01939002).
Sampling Method: Non-Probability Sample
Enrollment: 1208 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-01-20 (Actual)

PRIMARY OUTCOMES:
Safety as measured by the incidence proportion of SAEs | Up to 5 years
Safety as measured by the incidence rate of SAEs | Up to 5 years
Clinical no evidence of disease activity (NEDA) as measured by the proportion of participants with no relapses | Up to 5 years
Clinical NEDA as measured by the proportion of participants with no disability progression | Up to 5 years

SECONDARY OUTCOMES:
Prescription and utilization patterns as measured by prescribed dosing frequency | Up to 5 years
Prescription and utilization patterns as measured by duration of Plegridy use | Up to 5 years
Prescription and utilization patterns as measured by the primary reason for discontinuation of Plegridy | Up to 5 years
Relapse activity as measured by annualized relapse rate (ARR) | Up to 5 years
Relapse activity as measured by time to first relapse | Up to 5 years
Relapse activity as measured by the proportion of participants with relapse | Up to 5 years
Relapse activity as measured by the distribution of the number of relapses | Up to 5 years
Disability progression as measured by the proportion of participants with sustained progression for at least six months | Up to 5 years
  Disability progression measured by the Expanded Disability Status Scale (EDSS). The EDSS measures disability status on a scale ranging from 0 to 10, with higher scores indicating more disability. Scoring is based on measures of impairment in eight functional systems on examination by a neurologist. Participants with confirmed progression of disability in EDSS physical functional system scores will be defined as those who meet one of the following criteria: an increase of ≥ 1 point from baseline system score of ≥ 1 or an increase of ≥ 2 points from baseline system score of 0 in at least 2 physical functional systems, or an increase of ≥ 2 points from baseline system score of ≥ 1 or an increase of ≥ 3 points from baseline system score of 0 in any 1 physical functional system. Worsening must be confirmed on a subsequent examination using the same criterion in the same functional system(s) at least 6 months later.
Disability progression as measured by the time to sustained disability progression for at least six months | Up to 5 years
Incidence proportion of non-serious AEs leading to treatment discontinuation | Up to 5 years
Incidence rate of non-serious AEs leading to treatment discontinuation | Up to 5 years
Impact of the severity of FLS on the ability to successfully manage symptoms via prophylaxis as measured by the participant-reported FLS-VAS | Up to 5 years
Changes in FLS assessment and FLS-VAS over time | Baseline to 5 years
Changes in EuroQoL EQ-5D, 3-level (EQ-5D-3L) score over time | Baseline to 5 years
  The EQ-5D-3L is a standardized instrument for use as a measure of health outcome. It is a health questionnaire that consists of 2 pages - the EQ-5D descriptive system (page 2) and the EQ visual analogue scale (EQ VAS) (page 3). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.
Treatment adherence as measured by changes in adherence over time as reported in the treatment adherence questionnaires | Baseline to 5 years
  Where pen/syringe collection is locally allowed, treatment adherence will also be assessed by the proportion of used auto-injector pens/pre-filled syringes out of the total number of pens/syringes prescribed.
Frequency of MS-related and non-MS-related physician visits, specialists' visits, use of physiotherapy, hospitalizations and lengths of stay, and emergency room/department visits | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (142):
- United States (47):
  - Research Site, Homewood, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Berkeley, California
  - Research Site, California City, California
  - Research Site, Hanford, California
  - Research Site, Orange, California
  - Research Site, Basalt, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Delray Beach, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Schaumburg, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Des Moines, Iowa
  - Research Site, Iowa City, Iowa
  - Research Site, Louisville, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Scarborough, Maine
  - Research Site, Boston, Massachusetts
  - Research Site, Lexington, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Southfield, Michigan
  - Research Site, Golden Valley, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Great Falls, Montana
  - Research Site, Lebanon, New Hampshire
  - Research Site, Freehold, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Buffalo, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, Charlotte, North Carolina
  - Research Site, Hickory, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Port Royal, South Carolina
  - Research Site, Knoxville, Tennessee
  - Research Site, Bedford, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Virginia Beach, Virginia
  - Research Site, Milwaukee, Wisconsin
- Australia (6):
  - Research Site, Camperdown, New South Wales
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Auchenflower, Queensland
  - Research Site, Bedford Park, South Australia
  - Research Site, Fitzroy, Victoria
  - Research Site, Heidelberg, Victoria
- Austria (2):
  - Research Site, Linz
  - Research Site, Vienna
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Saint John, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Sydney, Nova Scotia
  - Research Site, Barrie, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Gatineau, Quebec
- Denmark (3):
  - Research Site, Esbjerg
  - Research site, Glostrup Municipality
  - Research Site, Sønderborg
- France (10):
  - Research Site, Nîmes, Gard
  - Research Site, Toulouse, Haute Garonne
  - Research Site, Montpellier, Herault
  - Research Site, Rennes, Ille Et Vilaine
  - Research Site, St-Malo, Ille Et Vilaine
  - Research Site, Le Mans, Sarthe
  - Research Site, La Seyne-sur-Mer, Var
  - Research Site, Poitiers, Vienne
  - Research Site, Mantes-la-Jolie, Yvelines
  - Research Site, Gonesse
- Germany (35):
  - Research Site, Aalen, Baden-Wurttemberg
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, Heidenheim, Baden-Wurttemberg
  - Research Site, Ladenburg, Baden-Wurttemberg
  - Research Site, Pforzheim, Baden-Wurttemberg
  - Research Site, Stuttgart, Baden-Wurttemberg
  - Research Site, Bamberg, Bavaria
  - Research Site, Munich, Bavaria
  - Research Site, Regensburg, Bavaria
  - Research Site, Rüdersdorf, Brandenburg
  - Research Site, Bad Homburg, Hesse
  - Research Site, Butzbach, Hesse
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Gelnhausen, Hesse
  - Research Site, Kassel, Hesse
  - Research Site, Göttingen, Lower Saxony
  - Research Site, Sande, Lower Saxony
  - Research Site, Stade, Lower Saxony
  - Research Site, Aachen, North Rhine-Westphalia
  - Research Site, Bonn, North Rhine-Westphalia
  - Research Site, Cologne, North Rhine-Westphalia
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Siegen, North Rhine-Westphalia
  - Research Site, Kandel, Rhineland-Palatinate
  - Research Site, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Research Site, Chemnitz, Saxony
  - Research Site, Leipzig, Saxony
  - Research Site, Itzehoe, Schleswig-Holstein
  - Research Site, Kiel, Schleswig-Holstein
  - Research Site, Altenburg, Thuringia
  - Research Site, Erfurt, Thuringia
  - Research Site, Jena, Thuringia
  - Research Site, Stadtroda, Thuringia
  - Research Site, Berlin
  - Research Site, Hamburg
- Research Site, Dublin, Ireland
- Italy (9):
  - Research Site, Bergamo
  - Research Site, Cagliari
  - Research Site, Catanzaro
  - Research Site, Florence
  - Research Site, Genova
  - Research Site, Messina
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Roma
- Netherlands (3):
  - Research Site, Blaricum
  - Research Site, Breda
  - Research Site, Hoorn
- Portugal (2):
  - Research Site, Guimarães
  - Research Site, Setúbal
- Spain (4):
  - Research Site, Cadiz
  - Research Site, Córdoba
  - Research Site, Málaga
  - Research Site, Seville
- Switzerland (4):
  - Research Site, Aarau
  - Research Site, Basel
  - Research Site, Bern
  - Research Site, Lucerne
- United Kingdom (8):
  - Research Site, Irvine, Ayrshire
  - Research Site, Truro, Cornwall
  - Research Site, London, Greater London
  - Research Site, Salford, Greater Manchester
  - Research Site, Inverness, Highland Region
  - Research Site, Leicester, Leicestershire
  - Research Site, Glasgow, Strathclyde
  - Research Site, Swansea

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on http://clinicalresearch.biogen.com/
URL: https://vivli.org/